CLINICAL TRIAL: NCT03740672
Title: Adherence to the Antiemesis National Comprehensive Cancer Network (NCCN) Guideline in Chinese Patients of Gynecologic Malignancies
Brief Title: Adherence to the Antiemesis National Comprehensive Cancer Network (NCCN) Guideline
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Lei Li (Other)
Responsible Party: Sponsor-Investigator, Lei Li, Professor, Peking Union Medical College Hospital
Organization: Peking Union Medical College Hospital (Other)
Other Study IDs: GO-CINV
Record Dates: First submitted 2018-11-10; First posted 2018-11-14 (Actual); Last update posted 2018-11-26 (Actual); Status verified 2018-11

CONDITIONS: Gynecologic Cancer; Chemotherapy-induced Nausea and Vomiting
MeSH Terms: conditions — Vomiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to investigate the adherence to the antiemesis NCCN guideline in Chinese patients of gynecologic malignancies, who are given chemotherapy treatment. The risk of chemotherapy induced nausea and vomiting (CINV) is calculated by the questionnaire supported by the website "CINV Risk Assessment" (http://www.riskcinv.org/).

ELIGIBILITY:
Inclusion Criteria:

* Good performance status
* Aged 18 years or older
* Signed an approved informed consents

Exclusion Criteria:

* Not meeting all of the inclusion criteria

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: All patients who are given chemotherapy treatment for gynecologic malignancies are included.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2018-11-22 (Actual); Primary Completion 2019-12-01 (Estimated); Study Completion 2019-12-01 (Estimated)

PRIMARY OUTCOMES:
risk of chemotherapy induced nausea and vomiting | One year
  The risk of chemotherapy induced nausea and vomiting is calculated by the questionnaire supported by the website "CINV Risk Assessment" (http://www.riskcinv.org/). The difference of patients adhered to and not to NCCN guideline is compared.

CONTACTS AND LOCATIONS:
Overall Officials: Lei Li, M.D., Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Lei Li, Beijing, Beijing Municipality, China